CLINICAL TRIAL: NCT00692406
Title: Neuroimaging Attentional Impairment During Abstinence
Acronym: SmokeAtt01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00007082
Record Dates: First submitted 2008-06-03; First posted 2008-06-06 (Estimated); Results first posted 2013-03-28 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2013-02

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Smokers not interested in quitting smoking (Experimental): Smokers were scanned 24 hours after quitting smoking, and scanned after smoking as usual.
  Interventions: Behavioral: Smoking Abstinence

INTERVENTIONS:
Behavioral: Smoking Abstinence — Smokers were scanned after having quitting smoking for 24 hours, and scanned after smoking as usual.

SUMMARY:
The broad objective of this proposal is to identify functional neuroanatomical correlates of impairments in sustained attention during smoking abstinence. We will measure changes in performance and regional blood oxygenation levels using fMRI while smokers and non-smokers complete a task designed to assess sustained attention-or the continuous monitoring of stimuli.

Our primary hypothesis is that smoking abstinence will result in impaired sustained attention accompanied by decreases in blood-oxygenation-level-dependent (BOLD) fMRI signal in regions associated with sustained attention including right fronto-parietal cortex, thalamus and reticular activation system. Abstinence may also result in performance-related increases in activation in brain regions associated with effortful processing including the anterior cingulate cortex. We also hypothesize that smokers during the satiated state will exhibit brain activity more similar to that of non-smokers.

In addition to task related brain responses, we will also measure changes in absolute regional cerebral blood flow (rCBF) and hypothesize that abstinence will result in significant decreases in regions associated with arousal (e.g., reticular activation system); information processing (e.g., thalamus); and emotional regulation (e.g., anterior cingulate cortex, prefrontal cortex).

DETAILED DESCRIPTION:
Following an extended training period in which performance will become stable, smokers will be tested in the 4 Tesla MRI scanner (GE LX NVi system) 24 hours after quitting smoking, and tested satiated, while non-smokers will be tested in the scanner once under normal conditions. This design will provide an assessment of how tobacco abstinence alters information processing.

Included smoker participants will smoke at least 10 cigarettes per day of a brand delivering at least 0.5 mg nicotine (by FTC method) for at least two years and have afternoon end tidal carbon monoxide (CO) concentrations of at least 10 ppm (confirming they are inhalers). Inclusion criteria for non-smoker participants is that they should have smoked less than 50 cigarettes in their lifetime, have not smoked or used any nicotine products during the last 6 months, and have afternoon end tidal CO of less than or equal to 5 ppm. In order to reduce variability and ensure comparable stimulus exposure, participants will be required to be right-handed, and have at least 20-30 corrected vision.

During a screening session, all aspects of the study will be described to subjects and informed consent will be acquired. Breath and saliva samples will be collected in order to verify smoking status; and paper-and-pencil measures of smoking history, nicotine dependence, and mood will be collected. Each subject will also complete a Brain Imaging and Analysis Center (BIAC) approved fMRI subject screening form. For females of child bearing potential, a blood sample will be taken for pregnancy testing. For all participants, a urine sample will be taken for illicit drug testing. Finally, each subject will be escorted to the hospital where they will view and be placed in a mock fMRI scanner for a short time in order to increase familiarity with study procedures. Subjects who meet all selection criteria will be scheduled for the remainder of sessions.

Participants will learn and practice a sustained attention task. The planned sustained attention task, called the rapid visual information processing task (RVIP) requires participants to identify series of three odd or three even numbers among a series of numbers presented one at a time on a computer monitor. A control task in which participants press a button when they see a '0' will also be practiced. Total task time is 15 minutes (practice version) and each participant will be required to complete as many as 8 practice versions or until 50% accuracy is achieved on two consecutive attempts. Training may require 2-8 visits but will not exceed 2 hours and 40 minutes in total duration. One practice version of the task will be conducted in the mock fMRI scanner.

Following the training period, smoker participants will complete two fMRI scans and non-smokers will complete one fMRI scan in which they will complete 1) undergo a five minute resting state BOLD scan, 2) two 12.5 minute versions of the RVIP and 3) a 12.5-minute 'cue-viewing' task in which they view pictures of people smoking. For the 'satiated' sessions, smoker participants will be instructed to smoke as usual before and after the session. For the 'abstinent' session, smoker participants will be required to quit smoking for 24 hours prior to the scan and 24 hours following the scan. Quitting will be verified using CO and salivary cotinine and nicotine levels collected at the time of the scan and a short session 24 hours after the scan. All smoker participants will be given information about quitting smoking for 48 hours and we will answer questions about quitting smoking. The order of the sessions-satiated first vs. abstinent first-will be randomly assigned.

One week after their second scan, participants will attend a 30-minute office visit in which they will complete questionnaires and the RVIP task.

ELIGIBILITY:
Inclusion Criteria:

1. smoked an average of 10 cigarettes per day for two years
2. a brand that delivers (by Federal Trade Commission rated yields) at least 0.5 mg nicotine
3. have an expired air carbon monoxide reading of at least 10 ppm.
4. be in general good health
5. Participants with controlled medical conditions (e.g., hypertension) will be considered if treatment is not thought to interfere with fMRI measures or potentially ameliorate smoking withdrawal symptoms

Exclusion Criteria:

1. Individuals with a major medical condition that would make participation unsafe (e.g., have pacemaker or other metallic implant),
2. uncomfortable (e.g., chronic pain),
3. confound results (e.g., psychiatric condition)
4. suffering from claustrophobia; abnormally afraid of closed-in places will be excluded from participation,
5. Current alcohol or drug abuse,
6. smokeless tobacco use, or use of nicotine replacement therapy or other smoking cessation treatment will also be a basis for exclusion and evaluated via a urine test.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2005-06; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis J McClernon, Ph.D, Principal Investigator — Duke UMC
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began on 6/23/05. We advertised in local newpapers, with flyers around Durham, and posting on dukeheatlh.org and dukesmoking.com. We recruited for this study until 11/08
Pre-assignment Details: If participants were excluded from the trial after enrollment it was due to inability to perform tasks, no shows to sessions, and or unsafe circumstances for the MRI sessions. Otherwise persons were lost to contact and/or decided to not participate anymore.
Groups:
- Smokers Not Interested in Quitting: Smokers were scanned twice, once following smoking as usual and once following 24 hrs smoking abstinence
Period: Overall Study
Arm/Group | Smokers Not Interested in Quitting
Started | 80 (Initially this group was assigned to quit smoking before the second scan.)
Completed | 23 (This group quit smoking before their second scan.)
Not Completed | 57
Not completed — PI dropped, bad data | 57

BASELINE CHARACTERISTICS:
Arm/Group | Smokers Not Interested in Quitting
Number analyzed (Participants) | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 80
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 31.4 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 37
Region of Enrollment [Number; unit: participants]
  United States | 80 (0)

OUTCOME MEASURES:

1. Primary Outcome: Percent Signal Change in fMRI BOLD Signal Between RVIP Task and Control Task in Inferior Frontal Gyri (IFG) During Sustained Attention Task on Satiated Day
Description: Percent signal change in BOLD (Blood Oxygenation Levels Dependent) signal between RVIP task and control task using functional Magnetic Resonance Imaging Signal in IFG following smoking as usual. Differences in brain activations were considered significant at p<.001.
Time Frame: 12.5 minutes of fMRI scanning following smoking as usual
Population: the reason the number of baseline participants does not match those analyzed is because of drop outs, screen fails, and excessive head motion during scanning.
Measure: Mean (Standard Deviation); unit: percentage of signal change
Groups:
- Smokers Not Interested in Quitting: Men and women ages 18-50 who smoke at least 10 cigarettes per day of a brand delivery at least 0.5 mg of nicotine for at least 2 years.
Arm/Group | Smokers Not Interested in Quitting
Number analyzed (Participants) | 19
percentage of signal change | -0.0023 (0.15467)
Statistical Analysis 1: Comparison: Smokers Not Interested in Quitting; Within group repeated measures design. Null hypothesis is that there will be no difference in percent signal change during active task relative to baseline; Test type: Superiority or Other; p < 0.001, ANOVA; Mean Difference (Final Values) = -0.0023

2. Primary Outcome: Percent Signal Change in fMRI BOLD Signal Between RVIP Task and Control Task in Inferior Frontal Gyri (IFG) During Sustained Attention Task on Abstinent Day
Description: Percent signal change in BOLD (Blood Oxygenation Levels Dependent) signal between RVIP task and control task using functional Magnetic Resonance Imaging Signal in IFG following not smoking for 24 hours. Differences in brain activations were considered significant at p<.001.
Time Frame: 12.5 minutes of fMRI scanning following 24 hrs smoking abstinence
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of signal change
Arm/Group | Smokers Not Interested in Quitting
Number analyzed (Participants) | 19
percentage of signal change | 0.1167 (0.19161)
Statistical Analysis 1: Comparison: Smokers Not Interested in Quitting; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.1167

3. Primary Outcome: Percent Signal Change in fMRI BOLD Signal Between RVIP Task and Control Task in Middle Frontal Gyri (MFG) During Sustained Attention Task on Satiated Day
Description: Percent signal change in BOLD (Blood Oxygenation Levels Dependent) signal between RVIP task and control task using functional Magnetic Resonance Imaging Signal in MFG following smoking as usual. Differences in brain activations were considered significant at p<.001.
Time Frame: 12.5 minutes of fMRI scanning following smoking as usual
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of signal change
Arm/Group | Smokers Not Interested in Quitting
Number analyzed (Participants) | 19
percentage of signal change | -0.0253 (0.22800)
Statistical Analysis 1: Comparison: Smokers Not Interested in Quitting; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA; Mean Difference (Final Values) = -0.0253

4. Primary Outcome: Percent Signal Change in fMRI BOLD Signal Between RVIP Task and Control Task in Middle Frontal Gyri (MFG) During Sustained Attention Task on Abstinent Day
Description: Percent signal change in BOLD (Blood Oxygenation Levels Dependent) signal between RVIP task and control task using functional Magnetic Resonance Imaging Signal in MFG following not smoking for 24 hours. Differences in brain activations were considered significant at p<.001.
Time Frame: 12.5 minutes of fMRI scanning following 24 hrs smoking abstinence
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of signal change
Arm/Group | Smokers Not Interested in Quitting
Number analyzed (Participants) | 19
percentage of signal change | 0.1432 (0.29593)
Statistical Analysis 1: Comparison: Smokers Not Interested in Quitting; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.1432

5. Primary Outcome: Percent Signal Change in fMRI BOLD Signal Between RVIP Task and Control Task in Angular Gyrus (AnG) During Sustained Attention Task on Satiated Day
Description: Percent signal change in BOLD (Blood Oxygenation Levels Dependent) signal using functional Magnetic Resonance Imaging Signal between RVIP task and control task in AnG following smoking as usual. Differences in brain activations were considered significant at p<.001.
Time Frame: 12.5 minutes of fMRI scanning following smoking as usual
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of signal change
Arm/Group | Smokers Not Interested in Quitting
Number analyzed (Participants) | 19
percentage of signal change | -0.0489 (0.08334)
Statistical Analysis 1: Comparison: Smokers Not Interested in Quitting; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA; Mean Difference (Final Values) = -0.0489

6. Primary Outcome: Percent Signal Change in fMRI BOLD Signal Between RVIP Task and Control Task in Angular Gyrus (AnG) During Sustained Attention Task on Abstinent Day
Description: Percent signal change in BOLD (Blood Oxygenation Levels Dependent) signal between RVIP task and control task using functional Magnetic Resonance Imaging Signal in AnG following not smoking for 24 hours. Differences in brain activations were considered significant at p<.001.
Time Frame: 12.5 minutes of fMRI scanning following 24 hrs smoking abstinence
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of signal change
Arm/Group | Smokers Not Interested in Quitting
Number analyzed (Participants) | 19
percentage of signal change | 0.0096 (0.15990)
Statistical Analysis 1: Comparison: Smokers Not Interested in Quitting; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.0096

7. Primary Outcome: Percent Signal Change in fMRI BOLD Signal Between RVIP Task and Control Task in Cuneus (Cun) During Sustained Attention Task on Satiated Day
Description: Percent signal change in BOLD (Blood Oxygenation Levels Dependent) signal between RVIP task and control task using functional Magnetic Resonance Imaging Signal in Cun following smoking as usual. Differences in brain activations were considered significant at p<.001.
Time Frame: 12.5 minutes of fMRI scanning following smoking as usual
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of signal change
Arm/Group | Smokers Not Interested in Quitting
Number analyzed (Participants) | 19
percentage of signal change | -0.0372 (0.17545)
Statistical Analysis 1: Comparison: Smokers Not Interested in Quitting; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA; Mean Difference (Final Values) = -0.0372

8. Primary Outcome: Percent Signal Change in fMRI BOLD Signal Between RVIP Task and Control Task in Cuneus (Cun) During Sustained Attention Task on Abstinent Day
Description: Percent signal change in BOLD (Blood Oxygenation Levels Dependent) signal using functional Magnetic Resonance Imaging Signal between RVIP task and control task in Cun following not smoking for 24 hours. Differences in brain activations were considered significant at p<.001.
Time Frame: 12.5 minutes of fMRI scanning following 24 hrs smoking abstinence
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: percentage of signal change
Arm/Group | Smokers Not Interested in Quitting
Number analyzed (Participants) | 19
percentage of signal change | 0.1210 (0.20106)
Statistical Analysis 1: Comparison: Smokers Not Interested in Quitting; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.1210

ADVERSE EVENTS:
Arm/Group | Smokers Not Interested in Quitting
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes